CLINICAL TRIAL: NCT05056064
Title: Efficacy of Swallowing Function After Early Postoperative Oral Exercise Among Patient With Oral Cavity Cancer Underwent Flap Reconstruction: A Randomized Controlled Trial
Brief Title: Efficacy of Swallowing Function After Early Postoperative Oral Exercise Among Patient With Oral Cavity Cancer Underwent Flap Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63222
Record Dates: First submitted 2021-09-05; First posted 2021-09-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-11

CONDITIONS: Oral Cavity Cancer
Keywords: Dysphagia; oral cancer; oral exercise
MeSH Terms: conditions — Mouth Neoplasms; Deglutition Disorders | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CA oral cavity (Experimental): Standard Treatment+Oral exercise
  Interventions: Other: Oral exercise
- control (No Intervention): Standard treatment

INTERVENTIONS:
Other: Oral exercise — exercise remain tongue
  Arms: CA oral cavity

SUMMARY:
Efficacy of swallowing function after early postoperative oral exercise among patient with oral cavity cancer underwent flap reconstruction: A randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* patient with CA tongue and tumor size 2 cm

Exclusion Criteria:

* previous treatment
* history of head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy swallowing function | 1 year
  Efficacy of swallowing function evaluate by Penetration-Aspiration scale by Rosenbek, this questionnaire classify patient for 8 score, from no entry of material into the larynx or trachea to material enters the trachea with no attempt to clear

CONTACTS AND LOCATIONS:
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No